CLINICAL TRIAL: NCT02143700
Title: Clinical Profile and Cognitive Status in Chronic Obstructive Pulmonary Disease's Patients
Brief Title: Cognitive Status in Chronic Obstructive Pulmonary Disease's Patients
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Assisstant professor, Universidad de Granada
Other Study IDs: DF0051UG
Record Dates: First submitted 2014-05-17; First posted 2014-05-21 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: exacerbation; cognitive; chronic obstructive pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Mental Status and Dementia Tests; Restraint, Physical; Observation

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Stable and exacerbated patients: Patients diagnosed of chronic obstructive pulmonary disease in a stable or exacerbated situation. Cognitive assessment of these patients will be performed.
  Interventions: Other: Cognitive assessment

INTERVENTIONS:
Other: Cognitive assessment — Patients are going to be assessed regarding the outcome measures
  Other Names: assessment; observation; evaluation

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a chronic condition involving an impairment in functionality and in the execution of activities of daily life. The hypothesis of this study is to examine the relationship between cognitive status and clinical profile (respiratory, sleep quality, nutritional status) in patients with chronic obstructive pulmonary disease in two different moments: exacerbation or stable situation.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease is a pathology with a systemic impact with a progressive evolution that is characterized by the presence of chronic airflow obstruction.

Patients with COPD may have problems with cognitive functioning, either globally or in single cognitive domains, such as information processing, attention and concentration, memory, executive functioning and self-regulation.

Several studies have determined the prevalence of cognitive impairment in COPD compared to healthy control subjects, reaching very high levels, 36% of COPD patients with mild cognitive impairment compared with 12 % non- COPD subjects.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease with exacerbation or stable.
* Signed written consent.
* Medical approval for inclusion

Exclusion Criteria:

* Heart disease.
* Neurological patients.
* Severe cognitive impairment in order not to complete the assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed of chronic obstructive pulmonary disease.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-08 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Cognitive impairment | Baseline
  The cognitive impairment will be measured using the Montreal Cognitive Assessment. The Montreal Cognitive Assessment is a test designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.

SECONDARY OUTCOMES:
Sleep quality | Baseline
  Participants are going to complete the Pittsburgh Quality of Sleep Index. This is a self-rating questionnaire with seven subscores that result in a global score between 0 and 21.
Activity monitoring | Baseline
  The accelerometer Armband is going to be used for activity monitoring. It measures the intensity of the activity during 12 hours.
Nutritional state | Baseline
  Mini Nutritional Assessment has been designed and validated to provide a single, rapid assessment of nutritional status in elderly patients in outpatient clinics, hospitals, and nursing homes. It is composed of simple measurements and brief questions that can be completed in about 10 min
Quality of life | Baseline
  Quality of life associated with health is going to be measured with two questionnaires: the EuroQol-5 questionnaire and the Health Questionnaire St. George
Cough | Baseline
  The Leicester Cough Questionnaire-acute is a validated cough-related health status questionnaire designed for patients with chronic cough.
Comorbidities | Baseline
  Comorbidities are going to be measured with the Charlson comorbidity index. The Charlson comorbidity index predicts the ten-year mortality for a patient who may have a range of comorbid conditions, such as heart disease, AIDS, or cancer (a total of 22 conditions). Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one.
Anxiety and depression | Baseline
  Patients are going to completed the Hospital Anxiety and Depression Scale composed of statements relevant to either generalized anxiety or depression.
Cognitive flexibility | Baseline
  The cognitive flexibility of patients is measured using the Trial Making Test. This test explores visual-conceptual and visual-motor tracking, and it is a frequently used neuropsychological test.
Forced vital capacity | Baseline
  Forced vital capacity is going to be measured with a spirometer as recommended by the American Thoracic Society
Forced expiratory volume in the first second | Baseline
  Forced expiratory volume in the first second is going to be measured with a spirometer as recommended by the American Thoracic Society

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy, Granada, Granada, Spain